CLINICAL TRIAL: NCT04908345
Title: Intraoperative Use Of Methadone In The Prevention of Postoperative Pain in Kidney Transplant Receptors
Brief Title: Methadone Anesthesia For Kidney Transplant Receptors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Felipe Chiodini Machado, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEFERENAL
Record Dates: First submitted 2021-05-20; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Renal Failure Chronic; Surgery
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Methadone; Fentanyl

STUDY DESIGN:
Intervention Model Description: Methadone x Fentanyl
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methadone (Experimental): Methadone 0,075mg/kg for induction and half of induction dose of boluses as needed during surgery
  Interventions: Drug: Methadone
- Fentanyl (Active Comparator): Fentanyl 3 mcg/kg for induction and half of induction dose of boluses as needed during surgery
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Methadone — Used at induction and during surgery
  Arms: Methadone
Drug: Fentanyl — Used at induction and during surgery
  Arms: Fentanyl

SUMMARY:
Intraoperative methadone or fentanyl will be administered to patients submitted to kidney transplant surgery. Postoperative pain, analgesic consumption and side effects will be evaluated

DETAILED DESCRIPTION:
Despite recent developments in postoperative pain control, many patients still experience moderate or severe pain after surgery. It is estimated that severe postoperative pain occurs in 20 to 40% of surgical procedures. With the development of kidney transplant services, a better study of the intraoperative analgesia used in this procedure and its impact on the postoperative is necessary. The management of postoperative pain in renal transplant recipients is essential to improve the quality of postoperative care, and may even impact the prognosis of the renal graft. One of the strategies to improve pain control in the perioperative period is the intraoperative use of intravenous methadone, given its pharmacokinetic profile. Methadone is an opioid agonist of µ receptors, it is also a Glutamate antagonist by blocking the N-methyl-D-aspartate (NMDA) receptor, and inhibits the reuptake of serotonin and norepinephrine. When administered in doses of 20 to 30mg, the analgesia generated by methadone can last from 24 to 36 hours. There is also evidence that the use of methadone in doses of 0.2 to 0.3 mg / kg is not associated with a higher incidence of side effects when compared to other opioids with short or intermediate duration of action, such as fentanyl, sufentanil and morphine. The aim of this study is to evaluate the effectiveness of using intraoperative methadone to reduce postoperative pain in patients undergoing kidney transplant surgery (recipients). Patients will be submitted to standardized general anesthesia, and the opioid used in anesthetic induction will be methadone or fentanyl with additional boluses if necessary. After extubation, Fentanyl will be installed in an intravenous analgesia pump controlled by the patient. Differences between groups regarding opioid consumption, pain scores, side effects and patient satisfaction will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* With indication for kidney transplant surgery
* Who sign the informed consent form

Exclusion Criteria:

* Patients who refuse to participate in the study
* Known allergy to any drug used in this protocol
* Presence of stage III or IV congestive heart failure
* Increase in QT interval on electrocardiogram (QT> 500 msec)
* Preemptive kidney transplantation (defined by transplantation in a patient who has not yet started kidney replacement therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Pain score 24h postoperatively | One day after surgery
  Reported pain in a scale of 0 (no pain) to 10 (maximum pain)
Pain score 48h postoperatively | Two days after surgery
  Reported pain in a scale of 0 (no pain) to 10 (maximum pain)
Pain score 72h postoperatively | Three days after surgery
  Reported pain in a scale of 0 (no pain) to 10 (maximum pain)
Analgesic use 24h postoperatively | One day after surgery
  Analgesic use after surgery
Analgesic use 48h postoperatively | Two days after surgery
  Analgesic use after surgery
Analgesic use 72h postoperatively | Three days after surgery
  Analgesic use after surgery

SECONDARY OUTCOMES:
Opioid-related side effects 24h postoperatively | One day after surgery
  Opioid-related side effects
Opioid-related side effects 48h postoperatively | Two days after surgery
  Opioid-related side effects
Opioid-related side effects 72h postoperatively | Three days after surgery
  Opioid-related side effects

CONTACTS AND LOCATIONS:
Overall Officials: Felipe C Machado, MD, PhD, Principal Investigator — USP
Locations (1):
- Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No